CLINICAL TRIAL: NCT06158386
Title: A Multicenter, Prospective, Single-arm Clinical Study on the Treatment of Refractory/Relapsed Follicular Lymphoma (R/RFL) With Chidamide Combined With Linperlisib
Brief Title: Chidamide Combined With Linperlisibon for the Treatment of Refractory/Relapsed Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Fujian Provincial Hospital (Other); Fujian Cancer Hospital (Other Government); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Jieyang People's Hospital (Other); Dongguan People's Hospital (Other Government); Huizhou Municipal Central Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Sun Yat-sen University (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-03
Record Dates: First submitted 2023-11-21; First posted 2023-12-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Follicular Lymphoma; Refractory B-Cell Lymphoma; Relapsed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with Linperlisib (Experimental)
  Interventions: Drug: Chidamide combined with Linperlisib

INTERVENTIONS:
Drug: Chidamide combined with Linperlisib — Specified dose on specified days: Cedarbenzamide (C) 20mg orally twice weekly, Limplica (L) 80mg once daily, 2 weeks on 2 weeks off, Repeat on day 28.

SUMMARY:
To observe the safety and efficacy of Chidamide combined with Linperlisib in the treatment of refractory and relapsed follicular lymphoma.

DETAILED DESCRIPTION:
This is a Phase 2, open-label clinical trial study that aims to evaluate the efficacy (eg. Complete response, Overall Survival, Progression Free Survival) and adverse effects of Chidamide combined with Linperlisib in the treatment of refractory and relapsed follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patients diagnosed with follicular lymphoma with grade 1-3a, have received at least second-line systemic treatment, and at least one of the first-line treatments includes anti-CD20 monoclonal antibody (anti-CD20 monoclonal antibody monotherapy or combined chemotherapy). If the latest histopathological diagnosis is more than 6 months, a lymph node or tissue puncture or biopsy (resection or coarse needle puncture) must be performed.
2. Age ≥18 years old, regardless of gender.
3. The estimated survival time is more than 3 months.
4. ECOG ≤ 2.
5. Be able to follow the requirements of the research plan.
6. The patients have at least one measurable lesion (any length of lymph node lesion > 1.5cm or any length of extranodal lesion > 1 cm) examined by computed tomography (CT)/ magnetic resonance imaging (MRI).
7. Be able to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. CNS involvement (current or previous).
2. Clinical evidence of transformation to a more aggressive subtype of lymphoma
3. Impaired bone marrow function: neutrophils < 1.5× 10*9/L, HB < 80 g/L, PLT < 75×10*9 /L, Impaired liver function, defined as serum total bilirubin > 1.5 x ULN or serum ALT and AST > 2.5x ULN, Patients with liver infiltration by lymphoma, AST and ALT > 5x ULN, Renal glomerular filtration rate (eGFR) < 30 ml/min.
4. PT INR>1.5ULN or APTT> 1.5 ULN, Serum amylase or lipase > 1ULN.
5. Patients with active infection of the human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV), if patients with HBV infection with HBsAg or hepatitis B core antibody (HBcAb) positive] but HBV DNA negative can be included, However, these patients need continuous antiviral treatment and HBV DNA PCR detection every cycle after enrollment.
6. Patients with CMV infection (IgM positive or CMV DNA was positive by PCR.)
7. Meet any of the following criteria related to visceral function: all kinds of clinically significant abnormal rhythm or conduction need clinical pre-diagnosis Hereditary QT interval syndrome or QTcF>480 msec or taking drugs that may cause Qt interval delay or torsade de pointes. A variety of clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, and coronary artery bypass grafting in the first 6 months of the group, with New York's cardiology (NYHA) classification of grade 3 or above. Left ventricular ejection fraction (LVEF )<40%, or uncontrolled blood pressure controlled by drugs (Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mgHg).
8. Have a history of stroke or intracranial hemorrhage within 6 months before drug administration for the first time.
9. Major surgery was performed within 4 weeks before enrollment.
10. Any PI3K inhibitor has been used before and the disease has progressed during the treatment period (within 6 months after the last use).
11. Received systemic anti-tumor therapy or radiotherapy within 4 weeks before enrollment.
12. The last time you participated in clinical trials of other drugs before enrollment was less than 2 weeks or the last time you used small molecular drugs (such as antibody drugs) was less than 4 weeks.
13. The patients received the transplantation of somatic hematopoietic stem cells within 3 months before enrollment.
14. Patients received allogeneic hematopoietic stem cell transplantation or had any active graft-versus-host disease within 6 months before drug administration.
15. Take a strong inducer or inhibitor of cytochrome P4503A4 (CYP3A4) within 2 weeks before the first drug administration (3 weeks for Hypericum perforatum)
16. Before the first drug administration, the toxic reaction of previous anti-tumor therapy has not recovered to ≤1 level (except alopecia).
17. Patients with uncontrolled systemic infection requiring intravenous antibiotic treatment.
18. Currently suffering from other primary tumors that need active treatment according to the guidelines.
19. Inability to take drugs orally, previous surgical history, or serious gastrointestinal diseases such as dysphagia and active gastric ulcer may affect the absorption of drugs.
20. Pregnant (serum pregnancy test results are positive) or lactating women
21. Any other diseases, abnormal metabolism, abnormal physical examination, or abnormal laboratory examination with significant clinical significance, according to the researcher's judgment, it is reasonable to suspect that the patient has a certain disease or state that is not suitable for using these two drugs, or it will affect the interpretation of the research results or put the patient in a high-risk situation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) | Up to 24 months
  CR was defined as the percentage of participants who achieved CR, using the Lugano criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 24 months
  Percentage of participants with best overall response of partial response (PR) and complete response (CR), using the Lugano criteria.
Progressive free survival (PFS) | Up to 24 months
  PFS was defined as the time from the date of treatment initiation to the date of first documentation of definitive disease progression (PD) or date of death from any cause, whichever occurs first.
Overall survival (OS) | Up to 24 months
  OS will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No